CLINICAL TRIAL: NCT05044234
Title: A Phase 2b, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety and Efficacy of Cedirogant (ABBV-157) in Adult Subjects With Moderate to Severe Psoriasis
Brief Title: A Study to Assess Adverse Events and Disease Activity With Cedirogant (ABBV-157) in Adult Participants With Moderate to Severe Psoriasis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company Decision
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M18-816
Record Dates: First submitted 2021-09-07; First posted 2021-09-14 (Actual); Results first posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Psoriasis
Keywords: Psoriasis; Plaque Psoriasis; Cedirogant; ABBV-157
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Placebo (Placebo Comparator): Participants received placebo capsules for cedirogant orally once daily (QD) for 16 weeks.
  Interventions: Drug: Placebo
- 75 mg Cedirogant (Experimental): Participants received 75 mg cedirogant orally once daily (QD) for 16 weeks.
  Interventions: Drug: Cedirogant
- 150 mg Cedirogant (Experimental): Participants received 150 mg cedirogant orally once daily (QD) for 16 weeks.
  Interventions: Drug: Cedirogant
- 375 mg Cedirogant (Placebo Comparator): Participants received 375 mg cedirogant orally once daily (QD) for 16 weeks.
  Interventions: Drug: Cedirogant

INTERVENTIONS:
Drug: Cedirogant — Capsule, Oral
  Other Names: ABBV-157
  Arms: 150 mg Cedirogant; 375 mg Cedirogant; 75 mg Cedirogant
Drug: Placebo — Capsule, Oral
  Arms: Placebo

SUMMARY:
Psoriasis is a chronic disease characterized by marked inflammation and thickening of the skin that results in thick, scaly skin plaques. This study assessed how safe and effective cedirogant (ABBV-157) was compared to placebo in adult participants with moderate to severe psoriasis. Efficacy and safety-related measurements assessed disease activity in participants with plaque psoriasis.

Cedirogant (ABBV-157) is an investigational drug being developed for the treatment of chronic plaque psoriasis. Participants were put into 1 of 4 groups, called treatment arms and each group received a different treatment. There was a 1 in 4 chance that participants were assigned to placebo.

Participants received oral daily doses of cedirogant or placebo capsules for 16 weeks.

There may have been a higher burden for participants in this study compared to usual standard of care. Participants attended regular visits per routine clinical practice. The effect of the treatment was checked by medical assessments, checking for side effects, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

- Participants with stable moderate to severe plaque psoriasis of at least 6 months duration and who are candidates for systemic therapy or phototherapy.

Exclusion Criteria:

* Primary non-responders to previous anti-interleukin (IL)-17 (e.g., secukinumab, ixekizumab, brodalumab), anti-IL-23 (e.g., guselkumab, tildrakizumab, risankizumab), or anti-IL-12/23 (e.g., ustekinumab) treatment for chronic plaque psoriasis.
* Diagnosis of erythrodermic psoriasis, generalized or localized pustular psoriasis, medication-induced or medication exacerbated psoriasis, or new onset guttate psoriasis or any other skin disease which may interfere with assessment of chronic plaque psoriasis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (53):
- United States (37):
  - UAB Department of Dermatology /ID# 238563, Birmingham, Alabama
  - Medical Dermatology Specialist /ID# 238518, Phoenix, Arizona
  - Arkansas Research Trials, LLC /ID# 238687, North Little Rock, Arkansas
  - Encino Research Center /ID# 245950, Encino, California
  - Velocity Clinical Research, Inc. /ID# 239536, North Hollywood, California
  - Medderm Associates /ID# 238834, San Diego, California
  - Lakes Research, LLC /ID# 238831, Miami, Florida
  - Florida International Rsrch cr /ID# 245959, Miami, Florida
  - Lenus Research & Medical Group /ID# 238695, Sweetwater, Florida
  - Advanced Clinical Research Institute /ID# 238697, Tampa, Florida
  - Clinical Research Trials of Florida, Inc. /ID# 238709, Tampa, Florida
  - ForCare Clinical Research /ID# 238856, Tampa, Florida
  - Cleaver Medical Group Dermatology - Dawsonville /ID# 246327, Dawsonville, Georgia
  - Marietta Dermatology Clinical Research /ID# 238679, Marietta, Georgia
  - Arlington Dermatology /ID# 238701, Rolling Meadows, Illinois
  - Dawes Fretzin, LLC /ID# 238704, Indianapolis, Indiana
  - Zel Skin & Laser Specialists - Edina /ID# 238714, Edina, Minnesota
  - Skin Specialists, PC /ID# 238514, Omaha, Nebraska
  - Forest Hills Dermatology Group /ID# 238708, Kew Gardens, New York
  - Buffalo Medical Group /ID# 239068, Williamsville, New York
  - Darst Dermatology /ID# 238677, Charlotte, North Carolina
  - Wilmington Dermatology Center /ID# 246445, Wilmington, North Carolina
  - Univ Hosp Cleveland /ID# 245953, Cleveland, Ohio
  - Dermatologists of Southwest Ohio, Inc /ID# 238939, Mason, Ohio
  - Oregon Dermatology and Research Center /ID# 238823, Portland, Oregon
  - University of Pittsburgh MC /ID# 246170, Pittsburgh, Pennsylvania
  - Clinical Partners, LLC /ID# 238620, Johnston, Rhode Island
  - Clinical Research Center of the Carolinas /ID# 238827, Charleston, South Carolina
  - Health Concepts /ID# 238510, Rapid City, South Dakota
  - Tennessee Clinical Research Center /ID# 238682, Nashville, Tennessee
  - Arlington Research Center, Inc /ID# 244171, Arlington, Texas
  - Orion Clinical Research /ID# 238619, Austin, Texas
  - Bellaire Dermatology Associates /ID# 247865, Bellaire, Texas
  - Center for Clinical Studies - Houston (Binz) /ID# 243700, Houston, Texas
  - Progressive Clinical Research /ID# 238565, San Antonio, Texas
  - Dermatology Specialists of Spokane /ID# 238809, Spokane, Washington
  - West Virginia Research /ID# 238517, Morgantown, West Virginia
- Canada (6):
  - Dr. Chih-ho Hong Medical Inc. /ID# 238864, Surrey, British Columbia
  - Wiseman Dermatology Research /ID# 238867, Winnipeg, Manitoba
  - SimcoDerm Medical and Surgical Dermatology Center /ID# 238861, Barrie, Ontario
  - Dr. Wei Jing Loo Medicine Prof /ID# 238865, London, Ontario
  - Lynderm Research Inc. /ID# 243199, Markham, Ontario
  - K. Papp Clinical Research /ID# 239695, Waterloo, Ontario
- Japan (10):
  - Nagoya City University Hospital /ID# 239286, Nagoya, Aichi-ken
  - Takagi Dermatology Clinic /ID# 239274, Obihiro-shi, Hokkaido
  - JR Sapporo Hospital /ID# 239277, Sapporo, Hokkaido
  - Mie University Hospital /ID# 239275, Tsu, Mie-ken
  - Okayama University Hospital /ID# 239285, Okayama, Okayama-ken
  - Kansai Medical University Hospital /ID# 239278, Hirakata-shi, Osaka
  - Hamamatsu University Hospital /ID# 239346, Hamamatsu, Shizuoka
  - The Jikei University Hospital /ID# 239319, Minato-ku, Tokyo
  - NTT Medical Center Tokyo /ID# 239287, Shinagawa-ku, Tokyo
  - Tokyo Medical University Hospital /ID# 239320, Shinjuku-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: ITT population: all randomized participants
Period: Overall Study
Arm/Group | Placebo | 75 mg Cedirogant | 150 mg Cedirogant | 375 mg Cedirogant
Started | 39 | 39 | 39 | 39
Completed | 10 | 13 | 12 | 12
Not Completed | 29 | 26 | 27 | 27
Not completed — Lost to Follow-up | 2 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 6 | 4 | 5 | 8
Not completed — Study terminated by Sponsor | 21 | 21 | 20 | 14
Not completed — Other, not specified | 0 | 0 | 1 | 2
Not completed — Delayed data entry | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT population: all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 75 mg Cedirogant | 150 mg Cedirogant | 375 mg Cedirogant | Total
Number analyzed (Participants) | 39 | 39 | 39 | 39 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (12.14) | 49.3 (10.13) | 45.3 (13.46) | 47.5 (12.11) | 46.6 (12.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 11 | 12 | 46
  Male | 30 | 25 | 28 | 27 | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15 | 6 | 36
  Not Hispanic or Latino | 32 | 31 | 24 | 33 | 120
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 9 | 12 | 11 | 8 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 2 | 3 | 1 | 1 | 7
  White | 27 | 24 | 26 | 30 | 107
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Psoriasis Area and Severity Index (PASI) Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.
  units on a scale | 20.11 (10.031) | 19.78 (8.698) | 20.58 (8.489) | 18.24 (8.048) | 19.68 (8.806)
Static Physicians Global Assessment (sPGA)--No. of participants with score of 3 or 4 at Baseline [Count of Participants; unit: Participants]
  Baseline score of 3 | 32 | 33 | 32 | 35 | 132
  Baseline score of 4 | 7 | 6 | 7 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving 75% Improvement in Psoriasis Area Severity Index (PASI) Score (PASI 75) at Week 16
Description: The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 75 is defined as at least a 75% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100.
Time Frame: Baseline, Week 16
Population: ITT population; the Observed Cases (OC) approach was used to handle missing data-- values for missing evaluations were not imputed, and a participant who had an evaluation on a scheduled visit was included in the OC analysis for that visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 75 mg Cedirogant | 150 mg Cedirogant | 375 mg Cedirogant
Number analyzed (Participants) | 12 | 14 | 13 | 12
percentage of participants | 0 [0.0 to 0.0] | 28.6 [4.9 to 52.2] | 7.7 [0.0 to 22.2] | 41.7 [13.8 to 69.6]

2. Secondary Outcome: Percentage of Participants Achieving a Static Physician Global Assessment (sPGA) Score of Clear or Almost Clear at Week 16
Description: The static Physicians Global Assessment (sPGA) is an assessment by the investigator of the overall disease severity at the time of evaluation. Erythema (E), induration (I), and desquamation (D) are scored on a 5-point scale ranging from 0 (none) to 4 (severe). The sPGA composite score ranges from 0 to 4 and is calculated as Clear (0) = 0 for all three; Almost clear (1) = mean >0, <1.5; Mild (2) = mean ≥1.5, <2.5; Moderate (3) = mean ≥2.5, <3.5; and Severe (4) = mean ≥3.5.
Time Frame: At Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 75 mg Cedirogant | 150 mg Cedirogant | 375 mg Cedirogant
Number analyzed (Participants) | 12 | 14 | 13 | 12
percentage of participants | 0 [0.0 to 0.0] | 21.4 [0.0 to 42.9] | 7.7 [0.0 to 22.2] | 33.3 [6.7 to 60.0]

3. Secondary Outcome: Percentage of Participants Achieving 50% Improvement in Psoriasis Area Severity Index (PASI) Score (PASI 50) at Week 16
Description: The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 50 is defined as at least a 50% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 75 mg Cedirogant | 150 mg Cedirogant | 375 mg Cedirogant
Number analyzed (Participants) | 12 | 14 | 13 | 12
percentage of participants | 8.3 [0.0 to 24.0] | 57.1 [31.2 to 83.1] | 38.5 [12.0 to 64.9] | 66.7 [40.0 to 93.3]

4. Secondary Outcome: Percentage of Participants Achieving 90% Improvement in Psoriasis Area Severity Index (PASI) Score (PASI 90) at Week 16
Description: The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 75 mg Cedirogant | 150 mg Cedirogant | 375 mg Cedirogant
Number analyzed (Participants) | 12 | 14 | 13 | 12
percentage of participants | 0 [0.0 to 0.0] | 14.3 [0.0 to 32.6] | 0 [0.0 to 0.0] | 33.3 [6.7 to 60.0]

5. Secondary Outcome: Percentage of Participants Achieving 100% Improvement in Psoriasis Area Severity Index (PASI) Score (PASI 100) at Week 16
Description: The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 100 is defined as at least a 100% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 75 mg Cedirogant | 150 mg Cedirogant | 375 mg Cedirogant
Number analyzed (Participants) | 12 | 14 | 13 | 12
percentage of participants | 0 [0.0 to 0.0] | 7.1 [0.0 to 20.6] | 0 [0.0 to 0.0] | 8.3 [0.0 to 24.0]

6. Secondary Outcome: Percentage of Participants Achieving Psoriasis Symptoms Scale (PSS) Total Score of 0 at Week 16 for Those With PSS >0 at Baseline
Description: The PSS is a 4-item patient-reported outcome (PRO) instrument that assesses the severity of psoriasis symptoms in participants with moderate to severe psoriasis. The symptoms included are: pain, redness, itching and burning from psoriasis. Current symptom severity is assessed as a daily diary, using a 5-point scale ranging from 0 (none) to 4 (very severe). The PSS total score is calculated by summing the scores of the questions and ranges from 0 to 16, where the higher the score, the greater the severity of psoriasis symptoms.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 75 mg Cedirogant | 150 mg Cedirogant | 375 mg Cedirogant
Number analyzed (Participants) | 11 | 13 | 12 | 11
percentage of participants | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 16.7 [0.0 to 37.8] | 18.2 [0.0 to 41.0]

7. Secondary Outcome: Percentage of Participants Achieving an Itch Numerical Rating Scale (NRS) ≥4-Point Improvement From Baseline at Week 16 for Participants With Itch NRS ≥4 at Baseline
Description: The itch NRS is an 11-point scale that participants completed to describe the intensity of their itch using a 24-hour recall period. The itch NRS asked the participants to: "Please rate your itching severity due to your psoriasis by circling the number that best describes your worst level of itching in the past 24 hours?" The itch NRS scale scores vary between 0, representing "no itching" and 10, representing "worst itch imaginable."
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 75 mg Cedirogant | 150 mg Cedirogant | 375 mg Cedirogant
Number analyzed (Participants) | 8 | 14 | 10 | 12
percentage of participants | 50.0 [15.4 to 84.6] | 42.9 [16.9 to 68.8] | 60.0 [29.6 to 90.4] | 66.7 [40.0 to 93.3]

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment to end of study; median time on follow-up was 109.0, 121.0, 130.0, and 103.0 days for the placebo, 75 mg cedirogant, 150 mg cedirogant and 375 mg cedirogant groups, respectively.
Description: TEAEs and SAEs were collected from first dose of study drug until 30 days after the last dose; mean time on treatment was 68.2 days for the placebo group, 71.6 days for the 75 mg cedirogant group, 71.2 days for the 150 mg cedirogant group, and 61.3 days for the 375 mg cedirogant group.
Arm/Group | Placebo | 75 mg Cedirogant | 150 mg Cedirogant | 375 mg Cedirogant
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39 | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 1/39 | 2/39
Other Adverse Events (participants affected / at risk) | 8/39 | 4/39 | 9/39 | 16/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=39) | 75 mg Cedirogant (N=39) | 150 mg Cedirogant (N=39) | 375 mg Cedirogant (N=39)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=39) | 75 mg Cedirogant (N=39) | 150 mg Cedirogant (N=39) | 375 mg Cedirogant (N=39)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
NASOPHARYNGITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
PSORIASIS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT05044234/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT05044234/SAP_001.pdf